CLINICAL TRIAL: NCT04068610
Title: A Phase Ib/II, Open-label, Multicenter Study of Novel Oncology Therapies in Combination With Chemotherapy and Bevacizumab as First-line Therapy in Metastatic Microsatellite-stable Colorectal Cancer (COLUMBIA-1)
Brief Title: COLUMBIA-1: Novel Oncology Therapies in Combination With Chemotherapy and Bevacizumab as First- Line Therapy in MSS-CRC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D910CC00001; 2019-000974-44 (EudraCT Number)
Record Dates: First submitted 2019-08-01; First posted 2019-08-28 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Microsatellite-stable Colorectal Cancer
Keywords: Microsatellite; colorectal; MSS-CRC; colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — durvalumab; Folfox protocol; Bevacizumab

STUDY DESIGN:
Intervention Model Description: The study is designed to concurrently evaluate potential novel combinations with clinical promise using a 2-part approach.
  Part 1 is a Phase 1b study of safety, and Part 2 is a Phase 2 study of efficacy and safety. The treatment regimens evaluated in Part 2 will depend on the evaluation of safety outcomes in Part 1.
  Following a screening period of up to 28 days, participants will be centrally assigned (Part 1) or randomized (Part 2) to one of the open study arms. In both study parts, study treatment may be administered until disease progression or any discontinuation criteria are met.
  In Part 2, experimental arms may be closed early based on futility from results of a planned interim analysis for each study arm. In both parts, new experimental arms consisting of FOLFOX and bevacizumab plus novel agent(s) may be added based on emerging nonclinical and clinical data via protocol amendment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab (Experimental): Participants in Part 1 safety run-in arm (S1) will receive intravenous (IV) infusions of FOLFOX (5-fluorouracil [5-FU]: 2400 mg/m^2 over 46-48 hours [Day 1 and 2 of every 14-day Cycle], oxaliplatin: 85 mg/m^2, folinic acid: 400 mg/m^2) and bevacizumab 5 mg/kg on Day 1 of every Cycle (14-day cycle) in combination with IV durvalumab 1500 mg every 4 weeks (Q4W) and IV oleclumab 3000 mg every 2 weeks (Q2W) till 4 doses (Cycle 4) then Q4W starting on Cycle 5 Day 1 until disease progression, unacceptable toxicity, withdrawal of participant consent, or another discontinuation criterion will be met.
  Interventions: Drug: Durvalumab; Drug: Oleclumab; Drug: FOLFOX; Drug: Bevacizumab
- Part 2 (C1): FOLFOX + Bevacizumab (Experimental): Participants in Part 2 control 1 arm (C1) will receive IV infusions of FOLFOX (5-FU: 2400 mg/m^2 over 46-48 hours [Day 1 and 2 of every 14-day Cycle], oxaliplatin: 85 mg/m^2, folinic acid: 400 mg/m^2) in combination with IV bevacizumab 5 mg/kg on Day 1 of every Cycle (14-day cycle) until disease progression, unacceptable toxicity, withdrawal of participant consent, or another discontinuation criterion will be met.
  Interventions: Drug: FOLFOX; Drug: Bevacizumab
- Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab (Experimental): Participants in Part 2 experimental 1 arm (E1) will receive IV infusions of FOLFOX (5-FU: 2400 mg/m^2 over 46-48 hours [Day 1 and 2 of every 14-day Cycle], oxaliplatin: 85 mg/m^2, folinic acid: 400 mg/m^2) and bevacizumab 5 mg/kg on Day 1 of every Cycle (14-day cycle) in combination with IV durvalumab 1500 mg Q4W and IV oleclumab 3000 mg Q2W till 4 doses (Cycle 4) then Q4W starting on Cycle 5 Day 1 until disease progression, unacceptable toxicity, withdrawal of participant consent, or another discontinuation criterion will be met.
  Interventions: Drug: Durvalumab; Drug: Oleclumab; Drug: FOLFOX; Drug: Bevacizumab

INTERVENTIONS:
Drug: Durvalumab — Participants will receive IV infusion of durvalumab as stated in arm description.
  Other Names: MEDI4736
  Arms: Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab; Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Drug: Oleclumab — Participants will receive IV infusion of oleclumab as stated in arm description.
  Other Names: MEDI9447
  Arms: Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab; Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Drug: FOLFOX — Participants will receive IV infusion of FOLFOX (5-FU, oxaliplatin, and folinic acid) as stated in arm description.
Drug: Bevacizumab — Participants will receive IV infusion of bevacizumab as stated in arm description.

SUMMARY:
COLUMBIA-1 is a Phase 1b/2 platform study to evaluate the safety and efficacy of standard of care (FOLFOX plus bevacizumab) alone and in combination with novel oncology therapies in first-line metastatic microsatellite-stable colorectal cancer (MSS-CRC).

DETAILED DESCRIPTION:
COLUMBIA-1 is a Phase 1b/2, open-label, multicenter, randomized, multidrug platform study to evaluate the safety and efficacy of standard of care (FOLFOX plus bevacizumab) in combination with novel oncology therapies in patients with first-line metastatic MSS-CRC. The study is designed to concurrently evaluate potential novel combinations with clinical promise using a 2-part approach. Part 1 is a Phase 1b study of safety, and Part 2 is a Phase 2 study of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally required authorization obtained from the participant/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Age ≥ 18 years at the time of screening.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Participants must have histologic documentation of advanced or metastatic CRC and: (a) A documented mutation test during screening and confirmed tumor locations from disease assessment for enrollment. (b) Participants must NOT have defective deoxyribonucleic acid (DNA) mismatch repair (MSI) as documented by testing. (c) Participants must not have received any prior systemic therapy for recurrent/metastatic disease (prior adjuvant chemotherapy or radio-chemotherapy is acceptable so long as progression was not within 6 months of completing the adjuvant regimen).
5. Participants must have at least one lesion that is measurable by RECIST v1.1 (Eisenhauer et al, 2009).
6. Participants must have adequate organ function.
7. Participants with medical conditions requiring systemic anticoagulation (eg, atrial fibrillation) are eligible provided that both of the following criteria are met: - The participant has an in-range International Normalized Ratio (INR) on a stable dose of oral anticoagulant or be on a stable dose of low molecular weight heparin. - The participant has no active bleeding or pathological condition that carries a high risk of bleeding.
8. Body weight >35 kg.
9. Adequate method of contraception per protocol.

Exclusion Criteria:

1. History of allogeneic organ transplantation.
2. Active or prior documented autoimmune disorders within the past 5 years.
3. History of venous thrombosis within the past 3 months.
4. Cardiovascular criteria: (a) Presence of acute coronary syndrome including myocardial infarction or unstable angina pectoris, other arterial thrombotic event including cerebrovascular accident or transient ischemic attack or stroke within the past 6 months. (b) New York Heart Association (NYHA) class II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or uncontrolled hypertension. (c) History of hypertensive crisis/hypertensive encephalopathy within the past 6 months.
5. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 ms.
6. No significant history of bleeding events or gastrointestinal perforation.
7. Uncontrolled intercurrent illness.
8. History of another primary malignancy except for: (a) Malignancy treated with curative intent and with no known active disease ≥ 5 years of low potential risk for recurrence. (b) Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease. (c) Adequately treated carcinoma in situ without evidence of disease.
9. History of active primary immunodeficiency.
10. Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus.
11. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
12. Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade > 1 from previous anticancer therapy.
13. History of leptomeningeal disease or cord compression.
14. Untreated central nervous system (CNS) metastases.
15. Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
16. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
17. Prior immunotherapy or anti-angiogenics.
18. Receipt of live attenuated vaccine within the past 30 days.
19. Major surgical procedure, open biopsy, or significant traumatic injury within the past 28 days.
20. Current or prior use of immunosuppressive medication within the past 14 days, with exceptions per protocol.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2026-11-24 (Estimated)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (11):
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, Ann Arbor, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Canton, Ohio
  - Research Site, Providence, Rhode Island
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Charlottesville, Virginia
- Australia (3):
  - Research Site, Clayton
  - Research Site, Heidelberg
  - Research Site, Melbourne
- Research Site, Toronto, Ontario, Canada
- France (2):
  - Research Site, Nantes
  - Research Site, Villejuif
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Segal NH, Tie J, Kopetz S, Ducreux M, Chen E, Dienstmann R, Hollebecque A, Reilley MJ, Elez E, Cosaert J, Cain J, Soo-Hoo Y, Hewson N, Cooper ZA, Kumar R, Tabernero J. COLUMBIA-1: a randomised study of durvalumab plus oleclumab in combination with chemotherapy and bevacizumab in metastatic microsatellite-stable colorectal cancer. Br J Cancer. 2024 Oct;131(6):1005-1013. doi: 10.1038/s41416-024-02796-3. Epub 2024 Jul 25. PMID 39048638
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910CC00001&attachmentIdentifier=96b0512e-b51a-43df-b987-a6328269f16a&fileName=D910CC00001_Clinical_Study_Protocol_Redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910CC00001&attachmentIdentifier=c859acb9-bfd6-4953-b4e2-74f82c4061e6&fileName=D910CC00001_Statistical_Analysis_Plan_Redacted.pdf&versionIdentifier=
- See also: CSR redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910CC00001&attachmentIdentifier=3b27ab74-79dc-4955-9155-d0f9fac2f93f&fileName=D910CC00001_Abbreviated_Study_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 61 participants were randomized in this study of which 59 participants received treatment.
Groups:
- Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab: Participants in Part 1 safety run-in arm (S1) received intravenous (IV) infusions of FOLFOX (5-fluorouracil [5-FU]: 2400 mg/m^2 over 46-48 hours [Day 1 and 2 of every 14-day Cycle], oxaliplatin: 85 mg/m^2, folinic acid: 400 mg/m^2) and bevacizumab 5 mg/kg on Day 1 of every Cycle (14-day cycle) in combination with IV durvalumab 1500 mg every 4 weeks (Q4W) and IV oleclumab 3000 mg every 2 weeks (Q2W) till 4 doses (Cycle 4) then Q4W starting on Cycle 5 Day 1 until disease progression, unacceptable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Part 2 (C1): FOLFOX + Bevacizumab: Participants in Part 2 control 1 arm (C1) received IV infusions of FOLFOX (5-FU: 2400 mg/m^2 over 46-48 hours [Day 1 and 2 of every 14-day Cycle], oxaliplatin: 85 mg/m^2, folinic acid: 400 mg/m^2) in combination with IV bevacizumab 5 mg/kg on Day 1 of every Cycle (14-day cycle) until disease progression, unacceptable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
- Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab: Participants in Part 2 experimental 1 arm (E1) received IV infusions of FOLFOX (5-FU: 2400 mg/m^2 over 46-48 hours [Day 1 and 2 of every 14-day Cycle], oxaliplatin: 85 mg/m^2, folinic acid: 400 mg/m^2) and bevacizumab 5 mg/kg on Day 1 of every Cycle (14-day cycle) in combination with IV durvalumab 1500 mg Q4W and IV oleclumab 3000 mg Q2W till 4 doses (Cycle 4) then Q4W starting on Cycle 5 Day 1 until disease progression, unacceptable toxicity, withdrawal of participant consent, or another discontinuation criterion was met.
Period: Overall Study
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Started | 7 | 26 | 26
Completed | 0 | 0 | 0
Not Completed | 7 | 26 | 26
Not completed — Death | 4 | 8 | 13
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 2
Not completed — Other | 3 | 12 | 11

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any study drugs and were analyzed according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab | Total
Number analyzed (Participants) | 7 | 26 | 26 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (12.4) | 55.5 (13.5) | 59.8 (12.5) | 57.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 11 | 21
  Male | 4 | 19 | 15 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 1 | 5
  Not Hispanic or Latino | 7 | 19 | 23 | 49
  Unknown or Not Reported | 0 | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 7 | 20 | 23 | 50
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) in Part 1
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 2.8 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
Participants
  Any TEAE | 7
  Any TESAE | 1

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in Part 1
Description: DLT: Any study drug related Grade (G)3 or higher toxicity including: any G3/G4 immune-mediated AE, any G3/4 noninfectious pneumonitis/colitis, transaminase elevation (TE) >8x upper limit of normal (ULN) or total bilirubin (TBL) >5xULN, increase in aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >=3xULN along with TBL >=2xULN, isolated liver TE >5 but =<8xULN or isolated TBL >3 but =<5xULN that does not downgrade to G1 or less within 14 days of onset, G3 nausea/vomiting/diarrhea that does not resolve to G2 or less within 3 days of maximal supportive care (MSC), G3/4 febrile neutropenia, G3/4 neutropenia not associated with fever/systemic infection, G4 anemia, G3 anemia with clinical sequelae/requires >2 units of red blood cells transfusion, thrombocytopenia (G4 >=7 days, G3 that did not improve by at least 1 grade within 7 days, G3/4 associated with G3/higher hemorrhage).
Time Frame: From Day 1 to 28 days after the first dose of novel oncology therapy (durvalumab and oleclumab)
Population: The DLT evaluable population included all participants in Part 1 safety run-in who received the full prescribed dose of durvalumab and ≥ 75% of the prescribed number of doses of FOLFOX plus bevacizumab and the other novel oncology therapy and completed the safety follow-up through the DLT evaluation period or experienced any DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
Participants | 0

3. Primary Outcome: Number of Participants With at Least 2-Grade Shift From Baseline to Worst Toxicity Grade in Clinical Laboratory Parameters in Part 1
Description: Number of participants with at least common terminology criteria for adverse events (CTCAE v5.0) 2-grade shift from baseline (last assessment prior to first dose) to worst toxicity grade in clinical laboratory parameters are reported. Clinical laboratory parameter analysis included hematology, clinical chemistry, coagulation, and urinalysis.
Time Frame: Baseline (Day 1) through 90 days after the last dose of study drug (approximately 2.8 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
Participants
  Hemoglobin (Hypo) | 1
  Lymphocytes (Hypo) | 2
  Neutrophils | 4
  Leukocytes (Hypo) | 3
  Activated Partial Thromboplastin Time | 1
  Albumin | 1
  Amylase | 2
  Bilirubin | 1
  Calcium Corrected (Hypo) | 1
  Creatine Kinase | 2
  Creatinine | 1
  Gamma Glutamyl Transferase | 1
  Glucose | 1
  Lipase | 5
  Magnesium (Hyper) | 1
  Magnesium (Hypo) | 1

4. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs in Part 1
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal finding in the vital sign parameters (body temperature, blood pressure, and pulse rate).
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 2.8 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
Participants
  Pyrexia | 2
  Temperature intolerance | 1
  Hypertension | 3

5. Primary Outcome: Percentage of Participants With Objective Response (OR) Per Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST v1.1) in Part 2
Description: The OR is defined as best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) based on RECIST v1.1 criteria. The CR is defined as disappearance of all target lesions (TLs) and non-target lesions (NTLs), normalization of tumor marker level, any pathological lymph nodes (target and non-target) must have reduction in short axis < 10 mm, and no new lesion. The PR is defined as at least a 30% decrease in the sum of the diameters (SoD) of TLs (compared to baseline) and no new lesions. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. In Part 2, randomization occurred between Day -8 and the same date as dosing.
Time Frame: Randomization through end of study (approximately 2.6 years)
Population: Intent-to-treat (ITT) population included participants who received any study drug and were analyzed according to the treatment group they were randomized to.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 26 | 26
Percentage of Participants | 46.2 [26.6 to 66.6] | 61.5 [40.6 to 79.8]
Statistical Analysis 1: Comparison: Part 2 (C1): FOLFOX + Bevacizumab vs Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab; Test type: Superiority; p = 0.3173, Cochran-Mantel-Haenszel; P-value for comparison of treatment arms obtained from stratified Cochran-Mantel-Haenszel test stratified by the location of the primary tumor; Odds Ratio (OR) = 1.8, 95% CI 2-sided [0.6 to 5.6]

6. Secondary Outcome: Percentage of Participants With OR Per RECIST v1.1 in Part 1
Description: The OR is defined as BOR of confirmed CR or confirmed PR based on RECIST v1.1 criteria. The CR is defined as disappearance of all TLs and NTLs, normalization of tumor marker level, any pathological lymph nodes (target and non-target) must have reduction in short axis < 10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the SoD of TLs (compared to baseline) and no new lesions. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation.
Time Frame: First dose (Day 1) through end of study (approximately 2.8 years)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
Percentage of Participants | 71.4 [29.0 to 96.3]

7. Secondary Outcome: Best Overall Response (BOR) Per RECIST v1.1 in Part 1
Description: BOR: best response including CR, PR, stable disease (SD), progressive disease (PD), and non-evaluable (NE) among all overall responses based on application of RECIST v1.1 to investigator assessments. CR: disappearance of all TLs and NTLs, normalization of tumor marker level, any pathological lymph nodes (target and non-target) must have reduction in short axis <10 mm, and no new lesions. PR: at least 30% decrease in the SoD of TL (compared to baseline) and no new NTL. Confirmation of CR and PR is required after 4 weeks. PD: at least a 20% increase in the SoDs of TLs, taking as reference the smallest sum on study, and an absolute increase of at least 5mm, or unequivocal progression of existing NTL, or new lesions. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD in at least 8 weeks from first dose of study drug. NE: either when no or only a subset of lesion measurements are made at an assessment. Number of participants with BOR are reported.
Time Frame: First dose (Day 1) through end of study (approximately 2.8 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
Participants
  CR | 0
  PR | 5
  SD >=8 weeks | 2
  PD | 0
  NE | 0

8. Secondary Outcome: Duration of Response (DoR) Per RECIST v1.1 in Part 1
Description: The DoR is defined as the time from the first documentation of a confirmed response (CR or PR) until the first documentation of PD or death due to any cause, whichever occurs first. The CR is defined as disappearance of all TLs and NTLs, normalization of tumor marker level, any pathological lymph nodes (target and non-target) must have reduction in short axis < 10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the SoD of TLs (compared to baseline) and no new lesion. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. The PD is defined as at least a 20% increase in the SoDs of TLs, taking as reference the smallest sum on study, and an absolute increase of at least 5 mm, or unequivocal progression of existing NTL, or new lesions. The DoR was analyzed using Kaplan-Meier method.
Time Frame: First dose (Day 1) through end of study (approximately 2.8 years)
Population: As-treated population included all participants who received any study drugs and were analyzed according to the treatment they actually received. The DoR was assessed for only those participants who had OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 5
Months | 6.0 [5.5 to NA] — Upper limit of 95% CI was not reached because an insufficient number of participants had DoR.

9. Secondary Outcome: Percentage of Participants With Disease Control (DC) Per RECIST v1.1 in Part 1
Description: The DC is defined as BOR of confirmed CR, confirmed PR, or stable disease (SD; maintained for ≥ 16 weeks) per RECIST v1.1. The CR is defined as disappearance of all TLs and NTLs, normalization of tumor marker level, any pathological lymph nodes (target and non-target) must have reduction in short axis < 10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the SoD of TLs (compared to baseline) and no new lesion. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Participants with SD will be included in the DC if they maintain SD for >= 16 weeks from start of treatment.
Time Frame: First dose (Day 1) through end of study (approximately 2.8 years)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
Percentage of Participants | 100 [59.0 to 100]

10. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST v1.1 in Part 1
Description: The PFS is defined as the time from assignment until the first documentation of PD or death due to any cause, whichever occurs first, regardless of whether the participant received subsequent anticancer therapy prior to progression. The PD is defined as at least a 20% increase in the SoDs of TLs, taking as reference the smallest sum on study, and an absolute increase of at least 5 mm, or unequivocal progression of existing NTL, or new lesions. The PFS was analyzed using the Kaplan-Meier method based on application of RECIST v1.1 to investigator assessments. Assignment occurred between Day -3 and -1.
Time Frame: Assignment through end of study (approximately 2.8 years)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
Months | 9.5 [7.8 to 18.2]

11. Secondary Outcome: Percentage of Participants With PFS at 12 Months (PFS-12) Per RECIST v1.1 in Part 1
Description: The PFS is defined as the time from assignment until the first documentation of PD or death due to any cause, whichever occurs first, regardless of whether the participant received subsequent anticancer therapy prior to progression. The PD is defined as at least a 20% increase in the SoDs of TLs, taking as reference the smallest sum on study, and an absolute increase of at least 5 mm, or unequivocal progression of existing NTL, or new lesions. The PFS was analyzed using Kaplan-Meier method based on application of RECIST v1.1 to investigator assessments. The percentage of participants progression free and alive at 12 months (PFS-12) are reported. Assignment occurred between Day -3 and -1.
Time Frame: Assignment through 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
Percentage of Participants | 28.6 [4.1 to 61.2]

12. Secondary Outcome: Overall Survival (OS) Per RECIST v1.1 in Part 1
Description: The OS is defined as the time from first dose until death due to any cause. The overall survival was analyzed using the Kaplan-Meier method based on application of RECIST v1.1 to investigator assessments.
Time Frame: First dose (Day 1) through end of study (approximately 2.8 years)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
Months | 30.1 [11.9 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed.

13. Secondary Outcome: Number of Participants With TEAEs and TESAEs in Part 2
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 2.6 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 26 | 26
Participants
  Any TEAE | 26 | 26
  Any TESAE | 7 | 12

14. Secondary Outcome: Number of Participants With at Least 2-Grade Shift From Baseline to Worst Toxicity Grade in Clinical Laboratory Parameters in Part 2
Description: Number of participants with at least CTCAE v5.0 2-grade shift from baseline (last assessment prior to first dose) to worst toxicity grade in clinical laboratory parameters are reported. Clinical laboratory parameter analysis included hematology, clinical chemistry, coagulation, and urinalysis.
Time Frame: Baseline (Day 1) through 90 days after the last dose of study drug (approximately 2.6 years)
Population: As-treated population included all participants who received any study drugs and were analyzed according to the treatment they actually received. Here, number analyzed (n) denotes number of participants analyzed for the specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 26 | 26
Participants
  Hemoglobin (Hypo) | 0 | 1
  Lymphocytes (Hyper) | 0 | 2
  Lymphocytes (Hypo) | 3 | 6
  Neutrophils | 7 | 8
  Platelets | 3 | 2
  Leukocytes (Hypo) | 2 | 4
  Activated Partial Thromboplastin Time | 5 | 5
  Albumin | 0 | 3
  Alkaline Phosphatase | 1 | 1
  Alanine Aminotransferase | 2 | 1
  Amylase | 7 | 3
  Aspartate Aminotransferase | 1 | 0
  Bilirubin | 1 | 1
  Calcium Corrected (Hypo) | 0 | 1
  Creatine Kinase: number analyzed (Participants) | 25 | 26
  Creatine Kinase | 2 | 3
  Creatinine | 2 | 2
  Gamma Glutamyl Transferase: number analyzed (Participants) | 26 | 25
  Gamma Glutamyl Transferase | 5 | 4
  Potassium (Hyper) | 0 | 2
  Potassium (Hypo) | 0 | 2
  Lipase | 12 | 15
  Magnesium (Hypo) | 0 | 1
  Sodium (Hypo) | 2 | 2

15. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs in Part 2
Description: as for outcome 4
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 2.6 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 26 | 26
Participants
  Pyrexia | 3 | 5
  Temperature intolerance | 5 | 5
  Hypertension | 4 | 4
  Hypotension | 1 | 1
  Supraventricular tachycardia | 1 | 0
  Ventricular tachycardia | 1 | 0

16. Secondary Outcome: BOR Per RECIST v1.1 in Part 2
Description: BOR: best response including CR, PR, SD, PD, NE among all overall responses based on application of RECIST v1.1 to investigator assessments. CR: disappearance of all TLs, NTLs, normalization of tumor marker level, any pathological lymph nodes (target, non-target) must have reduction in short axis <10 mm, no new lesions. PR: at least 30% decrease in the SoD of TL (compared to baseline) and no new NTL. Confirmation of CR, PR is required after 4 weeks. PD: at least a 20% increase in SoDs of TLs, taking as reference smallest sum on study, and an absolute increase of at least 5 mm, or unequivocal progression of existing NTL, or new lesions. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD in at least 8 weeks from first dose of study drug. NE: either when no or only a subset of lesion measurements are made at an assessment. Number of participants with BOR are reported. In Part 2, randomization occurred between Day -8 and the same date as dosing.
Time Frame: Randomization through end of study (approximately 2.6 years)
Population: The ITT population included participants who received any study drug and were analyzed according to the treatment group they were randomized to.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 26 | 26
Participants
  CR | 0 | 1
  PR | 12 | 15
  SD >=8 weeks | 11 | 6
  PD | 1 | 3
  NE | 2 | 1

17. Secondary Outcome: DoR Per RECIST v1.1 in Part 2
Description: The DoR is defined as the time from the first documentation of a confirmed response (CR or PR) until the first documentation of PD or death due to any cause, whichever occurs first. The CR is defined as disappearance of all TLs and NTLs, normalization of tumor marker level, any pathological lymph nodes (target and non-target) must have reduction in short axis < 10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the SoD of TLs (compared to baseline) and no new lesion. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. The PD is defined as at least a 20% increase in the SoDs of TLs, taking as reference the smallest sum on study, and an absolute increase of at least 5 mm, or unequivocal progression of existing NTL, or new lesions. The DoR was analyzed using Kaplan-Meier method. In Part 2, randomization occurred between Day -8 and the same date as dosing.
Time Frame: Randomization through end of study (approximately 2.6 years)
Population: The ITT population included participants who received any study drug and were analyzed according to the treatment group they were randomized to. The DoR was assessed for only those participants who had OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 12 | 16
Months | 7.7 [4.6 to 15.4] | 10.3 [5.8 to NA] — Upper limit of 95% CI was not reached because an insufficient number of participants had DoR.

18. Secondary Outcome: Percentage of Participants With DC Per RECIST v1.1 in Part 2
Description: The DC is defined as BOR of confirmed CR, confirmed PR, or SD (maintained for ≥ 16 weeks) per RECIST v1.1. The CR is defined as disappearance of all TLs and NTLs, normalization of tumor marker level, any pathological lymph nodes (target and non-target) must have reduction in short axis < 10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the SoD of TLs (compared to baseline) and no new lesion. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Participants with SD will be included in the DC if they maintain SD for >= 16 weeks from start of treatment. In Part 2, randomization occurred between Day -8 and the same date as dosing.
Time Frame: Randomization through end of study (approximately 2.6 years)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 26 | 26
Percentage of Participants | 88.5 [69.8 to 97.6] | 84.6 [65.1 to 95.6]

19. Secondary Outcome: PFS Per RECIST v1.1 in Part 2
Description: The PFS is defined as the time from randomization until the first documentation of PD or death due to any cause, whichever occurs first, regardless of whether the participant received subsequent anticancer therapy prior to progression. The PD is defined as at least a 20% increase in the SoDs of TLs, taking as reference the smallest sum on study, and an absolute increase of at least 5 mm, or unequivocal progression of existing NTL, or new lesions. The PFS was analyzed using the Kaplan-Meier method based on application of RECIST v1.1 to investigator assessments. In Part 2, randomization occurred between Day -8 and the same date as dosing.
Time Frame: Randomization through end of study (approximately 2.6 years)
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 26 | 26
Months | 11.1 [7.3 to 16.2] | 10.9 [6.9 to 15.1]

20. Secondary Outcome: Percentage of Participants With PFS at 12 Months (PFS-12) Per RECIST v1.1 in Part 2
Description: The PFS is defined as the time from randomization until the first documentation of PD or death due to any cause, whichever occurs first, regardless of whether the participant received subsequent anticancer therapy prior to progression. The PD is defined as at least a 20% increase in the SoDs of TLs, taking as reference the smallest sum on study, and an absolute increase of at least 5 mm, or unequivocal progression of existing NTL, or new lesions. The PFS was analyzed using Kaplan-Meier method based on application of RECIST v1.1 to investigator assessments. The percentage of participants progression free and alive at 12 months (PFS-12) are reported. In Part 2, randomization occurred between Day -8 and the same date as dosing.
Time Frame: Randomization through 12 months
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 26 | 26
Percentage of Participants | 38.6 [18.6 to 58.3] | 36.1 [17.1 to 55.5]

21. Secondary Outcome: OS Per RECIST v1.1 in Part 2
Description: The OS is defined as the time from randomization until death due to any cause. The overall survival was analyzed using the Kaplan-Meier method based on application of RECIST v1.1 to investigator assessments. In Part 2, randomization occurred between Day -8 and the same date as dosing.
Time Frame: Randomization through end of study (approximately 2.6 years)
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 26 | 26
Months | NA [20.6 to NA] — Median and upper limit of 95% CI could not be derived due to insufficient events being observed. | 22.4 [10.6 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed.

22. Secondary Outcome: Serum Concentrations of Durvalumab in Part 1 (S1) and Part 2 (E1)
Description: Serum concentrations of durvalumab collected over time in Part 1 (S1) and Part 2 (E1) are reported. The lower limit of quantification (LLOQ) for durvalumab was considered to be 50 ng/mL.
Time Frame: Part 1: Pre-dose on Day 1 of Cycle 1, 3, 7, 13; Part 2 (E1): Pre-dose on Day 1 of Cycle 1, 3, 7, 13, and 27
Population: Pharmacokinetic (PK) evaluable population included participants who received at least 1 dose of any study drug with at least 1 reportable PK concentration. Here, number of participants analyzed denotes those participants who were analyzed for this outcome measure. Number analyzed (n) denotes those participants who had adequate serum samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7 | 21
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 21
  Cycle 1 Day 1 | NA (NA) — Geometric mean and geometric CV% were not calculated as the concentration was below the LLOQ. | NA (NA) — Geometric mean and geometric CV% were not calculated as the concentration was below the LLOQ.
  Cycle 3 Day 1: number analyzed (Participants) | 6 | 18
  Cycle 3 Day 1 | 67980 (20.31) | 48600 (39.67)
  Cycle 7 Day 1: number analyzed (Participants) | 7 | 18
  Cycle 7 Day 1 | 112500 (28.63) | 97610 (46.56)
  Cycle 13 Day 1: number analyzed (Participants) | 4 | 14
  Cycle 13 Day 1 | 101500 (30.22) | 147000 (30.57)
  Cycle 27 Day 1: number analyzed (Participants) | 0 | 5
  Cycle 27 Day 1 |  | 120700 (29.83)

23. Secondary Outcome: Serum Concentrations of Oleclumab in Part 1 (S1) and Part 2 (E1)
Description: Serum concentrations of oleclumab collected over time in Part 1 (S1) and Part 2 (E1) are reported. The LLOQ for oleclumab was considered to be 1 µg/mL.
Time Frame: Part 1: Pre-dose on Day 1 of Cycle 1, 2, 7, and 13; Part 2 (E1): Pre-dose on Day 1 of Cycle 1, 2, 7, 13, and 27
Population: The PK evaluable population included participants who received at least 1 dose of any study drug with at least 1 reportable PK concentration. Here, number of participants analyzed denotes those participants who were analyzed for this outcome measure. Number analyzed (n) denotes those participants who had adequate serum samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7 | 22
µg/mL
  Cycle 1 Day 1 | NA (NA) — Geometric mean and geometric CV% were not calculated as the concentration was below the LLOQ. | NA (NA) — Geometric mean and geometric CV% were not calculated as the concentration was below the LLOQ.
  Cycle 2 Day 1: number analyzed (Participants) | 6 | 19
  Cycle 2 Day 1 | 111.2 (25.38) | 69.81 (199.1)
  Cycle 7 Day 1: number analyzed (Participants) | 7 | 19
  Cycle 7 Day 1 | 186.5 (53.45) | 159.8 (81.62)
  Cycle 13 Day 1: number analyzed (Participants) | 4 | 14
  Cycle 13 Day 1 | 146.7 (24.43) | 170.1 (35.77)
  Cycle 27 Day 1: number analyzed (Participants) | 0 | 5
  Cycle 27 Day 1 |  | 107.9 (30.42)

24. Secondary Outcome: Serum Concentrations of Bevacizumab in Part 1 (S1)
Description: Serum concentrations of bevacizumab collected over time in Part 1 (S1) are reported. The LLOQ for bevacizumab was considered to be 500 ng/mL.
Time Frame: Pre-dose on Day 1 of Cycle 1, 2, 7, 13, and 27
Population: The PK evaluable population included participants who received at least 1 dose of any study drug with at least 1 reportable PK concentration. Here, number analyzed denotes those participants who had adequate serum samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
ng/mL
  Cycle 1 Day 1 | NA (NA) — Geometric mean and geometric CV% were not calculated as the concentration was below the LLOQ.
  Cycle 2 Day 1: number analyzed (Participants) | 6
  Cycle 2 Day 1 | 36090 (16.55)
  Cycle 7 Day 1 | 73350 (39.94)
  Cycle 13 Day 1: number analyzed (Participants) | 5
  Cycle 13 Day 1 | 70370 (30.52)
  Cycle 27 Day 1: number analyzed (Participants) | 1
  Cycle 27 Day 1 | NA (NA) — Geometric mean and geometric CV% were not calculated as the concentration was below the LLOQ.

25. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) to Durvalumab in Part 1 (S1) and Part 2 (E1)
Description: Number of participants with positive ADA to durvalumab in Part 1 (S1) and Part 2 (E1) are reported.
Time Frame: Part 1: Pre-dose on Day(D)1 of Cycles(C)1 (baseline [BL]), 3, 7, 13, and 90 days post last dose of study drug (approximately 2.8 years); Part 2(E1):Pre-dose on D1 of C1 (BL), 3, 7, 13, 27, and 90 days post last dose of study drug (approximately 2.6 years)
Population: The ADA evaluable population included all participants who received at least 1 dose of any study drug, who have a non-missing baseline ADA result and at least 1 non-missing post-baseline ADA result. Number of participants analyzed (N) denotes the number of participants evaluated for this outcome measure. Number analyzed (n) denotes those participants who had adequate ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7 | 20
Participants
  ADA positive at baseline | 0 | 2
  ADA positive at Cycle 3 Day 1: number analyzed (Participants) | 7 | 16
  ADA positive at Cycle 3 Day 1 | 0 | 1
  ADA positive at Cycle 7 Day 1: number analyzed (Participants) | 7 | 18
  ADA positive at Cycle 7 Day 1 | 0 | 0
  ADA positive at Cycle 13 Day 1: number analyzed (Participants) | 4 | 13
  ADA positive at Cycle 13 Day 1 | 0 | 0
  ADA positive at Cycle 27 Day 1: number analyzed (Participants) | 0 | 5
  ADA positive at Cycle 27 Day 1 |  | 0
  ADA positive at 90 days post last dose: number analyzed (Participants) | 4 | 7
  ADA positive at 90 days post last dose | 0 | 0

26. Secondary Outcome: Number of Participants With Positive ADA to Oleclumab in Part 1 (S1) and Part 2 (E1)
Description: Number of participants with positive ADA to oleclumab in Part 1 (S1) and Part 2 (E1) are reported.
Time Frame: Part 1: Pre-dose on D1 of C1 (BL), 2, 7, 13, and 90 days post last dose of study drug (approximately 2.8 years); Part 2 (E1): Pre-dose on D1 of C1 (BL), 2, 7, 13, 27, and 90 days post last dose of study drug (approximately 2.6 years)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7 | 21
Participants
  ADA positive at baseline | 0 | 0
  ADA positive at Cycle 2 Day 1: number analyzed (Participants) | 6 | 17
  ADA positive at Cycle 2 Day 1 | 0 | 2
  ADA positive at Cycle 7 Day 1: number analyzed (Participants) | 7 | 18
  ADA positive at Cycle 7 Day 1 | 0 | 0
  ADA positive at Cycle 13 Day 1: number analyzed (Participants) | 4 | 13
  ADA positive at Cycle 13 Day 1 | 0 | 0
  ADA positive at Cycle 27 Day 1: number analyzed (Participants) | 0 | 5
  ADA positive at Cycle 27 Day 1 |  | 0
  ADA positive at 90 days post last dose: number analyzed (Participants) | 4 | 7
  ADA positive at 90 days post last dose | 0 | 0

27. Secondary Outcome: Number of Participants With Positive ADA to Bevacizumab in Part 1 (S1)
Description: Number of participants with positive ADA to bevacizumab in Part 1 (S1) are reported.
Time Frame: Pre-dose on D1 of C1 (BL), 2, 7, 13, 27, and 90 days post last dose of study drug (approximately 2.8 years)
Population: The ADA evaluable population included all participants who received at least 1 dose of any study drug, who have a non-missing baseline ADA result and at least 1 non-missing post-baseline ADA result. Here, number analyzed (n) denotes those participants who had adequate ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
Number analyzed (Participants) | 7
Participants
  ADA positive at baseline | 0
  ADA positive at Cycle 2 Day 1: number analyzed (Participants) | 6
  ADA positive at Cycle 2 Day 1 | 5
  ADA positive at Cycle 7 Day 1 | 7
  ADA positive at Cycle 13 Day 1: number analyzed (Participants) | 5
  ADA positive at Cycle 13 Day 1 | 5
  ADA positive at Cycle 27 Day 1: number analyzed (Participants) | 1
  ADA positive at Cycle 27 Day 1 | 1
  ADA positive at 90 days post last dose: number analyzed (Participants) | 4
  ADA positive at 90 days post last dose | 4

ADVERSE EVENTS:
Time Frame: Part 1: Day 1 through 90 days after the last dose of study drug (approximately 2.8 years); Part 2: Day 1 through 90 days after the last dose of study drug (approximately 2.6 years)
Description: As-treated population included all participants who received any study drugs and were analyzed according to the treatment they actually received.
Arm/Group | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab | Part 2 (C1): FOLFOX + Bevacizumab | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab
All-Cause Mortality (participants affected / at risk) | 4/7 | 8/26 | 13/26
Serious Adverse Events (participants affected / at risk) | 1/7 | 7/26 | 12/26
Other Adverse Events (participants affected / at risk) | 7/7 | 25/26 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab (N=7) | Part 2 (C1): FOLFOX + Bevacizumab (N=26) | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab (N=26)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (3)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (S1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab (N=7) | Part 2 (C1): FOLFOX + Bevacizumab (N=26) | Part 2 (E1): FOLFOX + Bevacizumab + Durvalumab + Oleclumab (N=26)
Amylase increased (Investigations) | 1 (1) | 5 (8) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 5 (5) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 3 (3) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 2 (2) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 4 (6) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 3 (4) | 4 (4)
Neutrophil count decreased (Investigations) | 4 (6) | 4 (6) | 4 (5)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 4 (7) | 3 (5)
Weight decreased (Investigations) | 2 (2) | 2 (2) | 2 (2)
Weight increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 5 (6) | 8 (9)
Dehydration (Metabolism and nutrition disorders) | 2 (4) | 3 (5) | 5 (5)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
Dysaesthesia (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (4) | 8 (8) | 4 (4)
Headache (Nervous system disorders) | 1 (2) | 5 (5) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 3 (3) | 5 (7)
Neurotoxicity (Nervous system disorders) | 0 (0) | 2 (4) | 3 (6)
Paraesthesia (Nervous system disorders) | 5 (6) | 7 (7) | 5 (7)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6) | 11 (18) | 10 (10)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 4 (4)
Irritability (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2) | 4 (6) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (6) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 2 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (5)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (4)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (5) | 4 (4) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 9 (11) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 12 (16) | 14 (19)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (3) | 2 (2) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 13 (16) | 12 (12)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 3 (5)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Rectal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 5 (5) | 8 (9)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 6 (13)
Asthenia (General disorders) | 0 (0) | 2 (3) | 4 (7)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0)
Crepitations (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (7) | 10 (16) | 11 (12)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (10) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 3 (3) | 1 (3)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 3 (3) | 5 (11)
Temperature intolerance (General disorders) | 1 (1) | 5 (5) | 5 (5)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (4) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (5)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 3 (4)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (4) | 2 (2)

LIMITATIONS AND CAVEATS:
The data cut-off for the study was October 2022. The decision was made to end recruitment for the study because superior efficacy was not observed for the novel study drug combinations under investigation. For patient that were benefiting from the treatment the study remained active for them to continue receiving treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT04068610/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT04068610/SAP_001.pdf